CLINICAL TRIAL: NCT03577340
Title: Development and Validation of Performance Metrics for Cardiac Device
Brief Title: Development and Validation of Performance Metrics for Cardiac Device Implant Procedures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Archana Rao, Consultant Cardiologist, Liverpool Heart and Chest Hospital NHS Foundation Trust
Other Study IDs: 1189
Record Dates: First submitted 2018-06-22; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Educational Problems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Novices: Novices: Trainee cardiologists implanting cardiac devices as per guidelines under supervision
  Interventions: Other: implant of cardiac device as per guidelines
- Experts: Experts: Device implanting cardiologists implanting cardiac devices as per guidelines
  Interventions: Other: implant of cardiac device as per guidelines

INTERVENTIONS:
Other: implant of cardiac device as per guidelines — Observation of performance to validate matrix

SUMMARY:
Cardiac Device implantation includes implantation of pacemakers, implantable defibrillators and Cardiac resynchronisation Therapy (CRT) devices. These are well-established treatments for selected with heart rhythm abnormalities and heart failure.

In the past, trainee doctors had the opportunity to perform many procedures and learn on the patient. This is no longer the case due to a change in training schedules and working times as well as patient safety mandates. Progression based training with the use of simulators has been proven to be effective in training and in order to use this methodology, the procedure needs to be well defined.

Despite its worldwide adoption, a standardized procedure has never been defined in detail and agreed upon and the cardiac device implant technique varies with the operator.

The purpose of the research is to establish the metrics (operational definitions) necessary to characterize a reference Cardiac Device implant procedure.

DETAILED DESCRIPTION:
The purpose of the research is to establish the metrics (operational definitions) necessary to characterize a reference Cardiac Device implant procedure, to seek consensus from experienced device implanters on the appropriateness of the steps as well as errors identified, and to determine if such validated performance metrics are a valid assessment tool with the ability to discriminate between the performances of experienced and novice implanters.

These validated metrics will potentially serve as an educational and training tool to improve and quality assure Cardiac device implant training.

The steps involved in characterising a reference procedure are as follows:

1. Define the implant procedure in quantifiable steps (already performed)
2. Seek consensus and agreement by an independent panel on the steps (already done).
3. Video record routinely performed device implants by experienced and novice physicians.
4. Reviewing and scoring the video recorded procedures to verify that the metrics distinguish between a novice and an expert cardiac device performance.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for a cardiac device implant as per current European Society of Cardiology guidelines.

Exclusion Criteria:

Patient< 18 y of age. Patients unable to provide informed written consent for the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational and educational study only. Cardiac device implants routinely performed in clinical practice will be video-recorded.
  The procedures will be scheduled as per normal and the clinical pathway and management of the patient and the operator will remain unchanged.
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the comparison of the intra-operative performance of novices versus experts | 6 months
  The primary analysis will compare the intra-operative performance of novices versus experts.
  The three experienced cardiac device implanters will test the consented metrics by reviewing and scoring the video recorded procedures to verify that the metrics distinguish between a novice and an expert cardiac device performance. IRR will be considered to be acceptable if it is ≥ 0.8 The primary analysis will compare the intra-operative performance of novices versus experts.
  The three experienced cardiac device implanters will test the consented metrics by reviewing and scoring the video recorded procedures to verify that the metrics distinguish between a novice and an expert cardiac device performance. IRR will be considered to be acceptable if it is ≥ 0.8

IPD SHARING:
Plan to Share IPD: Yes
Presentation at national and international meetings
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12 months
Access Criteria: as above